CLINICAL TRIAL: NCT07007481
Title: SOOTH-ED: Purrble's Soothing Touch for Eating Disorders and Autism
Brief Title: Purrble's Soothing Touch for Eating Disorders and Autism
Acronym: SOOTH-ED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 333898; 10.17605/OSF.IO/4UKFW (Other: OSF)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders; Autism Spectrum Disorder
Keywords: Eating Disorders; Autism; Sensory Porcessing; Emotion Regulation; Purrble
MeSH Terms: conditions — Feeding and Eating Disorders; Autism Spectrum Disorder; Autistic Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Purrble) (Experimental): Participants in this group will be provided with the Purrble device, while waitlisted for eating disorder treatment.
  Interventions: Device: Purrble
- Control Group (No Intervention): The control condition will be waitlist as usual. Participants in this arm will not receive the Purrble intervention and will serve as a reference group for comparison.

INTERVENTIONS:
Device: Purrble — The intervention takes the form of an interactive plush toy, which was co-designed with children to support in-the-moment soothing. The device is framed as an anxious creature, in need of care and attention when it feels distressed. This distress is indicated by a simulated heartbeat using embedded electronics to produce vibration patterns of i) frantic and anxious, to ii) slow, steady and relaxed. When held, the device emits a frantic heartbeat which can be slowed by stroking movements registered by embedded sensors. Once the device has been "soothed" for long enough, the heartbeat transitions into a purring vibration indicating a relaxed state. This transition can be achieved in under 1 minute but is dependent on the device-human interaction.
  Arms: Intervention Group (Purrble)

SUMMARY:
The purpose of this study is to explore the potential therapeutic benefits of the Purrble intervention, a tangible device designed to assist with in-situ emotion regulation, for individuals on the South London and Maudsley NHS Trust (SLaM) Eating Disorders outpatient service waiting list. By examining its effects on emotion regulation, sensory sensitivity, depression, anxiety, and motivation for treatment engagement, the study seeks to offer empirical evidence on the efficacy of the Purrble as a supportive tool while patients are on the waiting list for formal outpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled on the South London and Maudsley NHS Foundation Trust (SLaM) Eating Disorders Outpatient Service waiting list
* Confirmed diagnosis of an ED.
* Participants aged 18 and above.
* Willing to commit to the duration of the study and provide informed consent.

Exclusion Criteria:

* Individuals currently dealing with substance abuse issues.
* Individuals with active psychosis.
* Individuals currently experiencing high suicidality or deemed to be at a high risk of self-harm.
* Individuals currently undergoing a separate ED treatment.
* Individuals who have previously been exposed to the Purrble intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale DERS-8 | From enrollment to the end of intervention at 4 weeks
  DERS-8 is a unidimensional measure of emotion regulation difficulties in adolescents and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Tchantura, PhD, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing may be considered in the future upon request and pending appropriate approvals.

REFERENCES:
- [Background] Slovak P, Ford BQ, Widen S, Dauden Roquet C, Theofanopoulou N, Gross JJ, Hankin B, Klasnja P. An In Situ, Child-Led Intervention to Promote Emotion Regulation Competence in Middle Childhood: Protocol for an Exploratory Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 9;10(11):e28914. doi: 10.2196/28914. PMID 34751666
- [Background] Kinnaird E, Dandil Y, Li Z, Smith K, Pimblett C, Agbalaya R, Stewart C, Tchanturia K. Pragmatic Sensory Screening in Anorexia Nervosa and Associations with Autistic Traits. J Clin Med. 2020 Apr 20;9(4):1182. doi: 10.3390/jcm9041182. PMID 32326069
- [Background] Brockmeyer T, Skunde M, Wu M, Bresslein E, Rudofsky G, Herzog W, Friederich HC. Difficulties in emotion regulation across the spectrum of eating disorders. Compr Psychiatry. 2014 Apr;55(3):565-71. doi: 10.1016/j.comppsych.2013.12.001. Epub 2013 Dec 7. PMID 24411653

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT07007481/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT07007481/ICF_001.pdf